CLINICAL TRIAL: NCT04057976
Title: The Accuracy of Advanced Probabilistic Diffusion Tensor Tractography (DTT) for the Pre-operative Identification of Facial Nerve Position in Patients With Extrameatal Vestibular Schwannomas.
Brief Title: Use of DTT to Define Facial Nerve Position in Vestibular Schwannomas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 226479
Record Dates: First submitted 2019-07-11; First posted 2019-08-15 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2024-10

CONDITIONS: Vestibular Schwannoma
MeSH Terms: conditions — Neuroma, Acoustic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients having pre-operative DTT prior to surgery (Experimental): All patients in this study will undergo DTT as part of a pre-operative MRI.
  Interventions: Diagnostic Test: Probabilistic diffusion tensor tractography

INTERVENTIONS:
Diagnostic Test: Probabilistic diffusion tensor tractography — Patients enrolled in this study will undergo probabilistic diffusion tensor tractography (additional MRI sequence) preoperatively in order to determine whether this it is possible to determine the course of the facial nerve.

SUMMARY:
Vestibular schwannomas (VS) arise from the vestibulocochlear (hearing and balance) nerve, located at the base of the brain. Although benign, VS can enlarge over time, resulting in debilitating symptoms; therefore, surgical removal is frequently offered. One significant risk of surgery is inadvertent injury to the facial nerve, which lies adjacent to the vestibulocochlear nerve. Currently, the nerve's course is only revealed during surgical dissection and injury can cause permanent facial weakness. It would therefore be useful for the surgeon to know the course of the nerve before operating. To this end, a new MRI technique known as probabilistic diffusion tensor tractography (DTT) has shown potential in revealing the course of the facial nerve pre-operatively. However, its clinical reliability remains uncertain.

This study aims to investigate the reliability of DTT in identifying the course of the facial nerve preoperatively in patients undergoing surgery for VS.

The future benefit would be to enable surgeons to operate with more confidence and potentially reduce the chance of nerve injury.

The study will recruit adult patients due to have surgery for VS. The only change to the participants' clinical pathways will be the addition of a DTT sequence to their pre-operative MRI scans (increasing scanning time by approximately 10 minutes).

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE Vestibular schwannomas (VS) are peripheral nerve sheath tumours arising from the vestibulocochlear nerve, which emerges from the brainstem at the base of the brain and enters the structures of the inner ear via a small bony canal within the skull (internal auditory meatus). VS account for 8% (Johnson J et al.) of intracranial tumours and, although benign, these tumours can grow resulting in several potentially debilitating symptoms, including hearing loss, vertigo, tinnitus, facial paralysis and meningitis. Furthermore, large tumours may cause compression on the brainstem, which can, in some cases, have life-threatening consequences (Johnson J et al.). Therefore, patients diagnosed with larger tumours (>1.5cm extrameatal component) are frequently offered surgical resection (as opposed to conservative management or stereotactic radiosurgery). As surgical techniques have improved, the goal of surgery has broadened to include not only tumour removal, but also preservation of the function of the nerves involved by VS. In particular, surgical resection aims to preserve the function of the facial nerve, responsible for innervating the muscles of facial expression, and which runs alongside the vestibulocochlear nerve and is frequently displaced and flattened by VS. Given its juxtaposition, the facial nerve is at high risk of injury during surgery. Injury to the facial nerve (and consequent debilitating facial weakness or paralysis) is a serious potential risk of vestibular schwannoma (VS) surgery. However, at present, the only means of avoiding nerve injury involves a combination of meticulous surgical technique and the use of a facial nerve monitor (a device that can detect activity within the facial muscles when stimulated by a surgeon-held probe); however, despite this, facial nerve injury may still occur. Indeed, until the surgeon begins operating, the course of the facial nerve is unknown. In a large series (>1000 surgical cases) by Sampath et al., the position of the facial nerve position was found most commonly on the anterior middle portion of the tumour; however, in a smaller proportion of cases, the nerve lay in 1 of 7 additional locations (Sampath et al.). Therefore, it follows that preoperative detection and identification of the course of the facial nerve would be extremely useful to guide surgery and reduce the potential risk of neuronal injury.

There now exists a potential means of non-invasively identifying the course of the facial nerve using advanced applications of magnetic resonance imaging (MRI). This involves utilising a technique known as diffusion tensor tractography (DTT), which has the capacity to detect the direction (vector) of diffusivity in a particular volume of tissue (voxel) (Mukherjee et al.). This data can be subsequently used to reveal structures, such as nerve fibre tracts, that are arranged along particular vectors, enabling them to be differentiated from surrounding tissue (Cauley et al.). This cannot be achieved using standard MRI sequences, in which the flattened nerve often becomes indistinguishable from the adjacent VS. Fortunately, as MRI represents the current means of diagnosing and characterising VS, adding an additional DTT sequence to a patient's scan does not represent a significant burden (only approximately 10 additional minutes of scanning time to acquire the DTT data).

Several groups (Choi et al., Taoka et al., Gerganov et al., Zhang et al. and Song et al.) have used DTT to delineate the course of the facial nerve in patients with VS and the majority have reported high success rates (>90% agreement with operative findings). However, many of these studies employed 'deterministic' DTT, which has drawbacks that limit its reliability in the setting of small fibre tracts with complex geometry. In particular, it is unable to accurately track fibres that cross, split or merge because the technique assumes that adjacent voxels have similar vectors. In order to overcome these limitations, we propose using the newer 'probabilistic' DTT technique that calculates a vector for each voxel analysed. It therefore has the capacity to account for complex geometries, such as those encountered in the facial nerve, particularly where its course is heavily distorted by tumour tissue. Zolal et al. used this technique in 21 patients with VS, resulting in an agreement rate of 81% for the position of the facial nerve and 33% for the cochlear nerve (Zolal et al.). However, there is an ongoing need for further studies in this area.

This project seeks to clarify the accuracy, reproducibility and practicality of probabilistic DTT in locating the facial nerve pre-operatively. If the technique proves accurate, it will potentially help with pre-operative planning and avoidance of facial nerve injury during VS surgery. Additionally the project seeks to clarify associated practical issues; in particular, the inter-observer/intra-observer variability (i.e. whether the reading radiologists agree with each other and themselves when analysing DTT images), whether the facial nerve position can be partially inferred on conventional sequences (comparing this with DTT) and whether adjacent nerves (such as the vestibulocochlear nerve) can be identified, which may further help with surgical preoperative planning.

HYPOTHESIS:

It is hypothesised that preoperative advanced probabilistic diffusion tensor tractography (DTT) will accurately demonstrate the position of the facial nerve relative to extrameatal portion of a vestibular schwannoma. It is proposed that the accuracy will be superior to previous studies in which deterministic DTT has been used to demonstrate the position of the facial nerve. This pre-operative mapping has the potential to decrease the rates of facial nerve injury during vestibular schwannoma surgery and allow for increased resection of the tumour.

STUDY DESIGN:

Prospective cohort observational study.

For study eligibility and outcome measures, please see the relevant sections.

IMAGE ANALYSIS

MRI In addition to standard imaging assessment, further image analysis will be performed offline using MRTrix 3.0 (www.mrtrix.org) in tensor probabililty mode. The presence of one or more cranial nerve tracts will be determined by their consistent depiction following their systematic interrogation with varying anisotropy thresholds. There will be a qualitative assessment of cranial nerve position will be achieved by dividing the circumference of the extrameatal vestibular schwannoma into segments.The assessment will be performed by two observers.

Reference standard:

The position of the facial nerve with respect to the extrameatal portion of the vestibular schwannoma will be assessed at surgery will be achieved by dividing the circumference of the extrameatal vestibular schwannoma into multiple segments in the same manner as above. This assessment will be made independently of the results of the pre-operative probabilistic DTT (the neurosurgeon recording the data will be blinded to the DTT findings).

STATISTICAL CONSIDERATIONS

Sample size calculation:

Power calculation based upon a sample size of 32, assuming a true kappa coefficient of 0.9; the 95% confidence interval will have a width of 0.26 (0.77 - 1.03). The number (32) also reflects the number of cases that we expect to recruit over a 2-3 year period.

ELIGIBILITY:
Inclusion Criteria:

* The capacity to understand the patient information sheet and the ability to provide written informed consent
* >1.5cm extrameatal tumor determined to represent a vestibular schwannoma by preoperative imaging
* HB grade I or II preoperatively

Exclusion Criteria:

* Patients not meeting the above inclusion criteria
* Standard contraindications to MRI
* Previous cranial radiotherapy or previous surgery to the cerebellopontine angle cistern or IAM

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-06-27 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Accuracy of probabilistic diffusion tensor tractography (DTT) | 4 years
  To assess the accuracy of pre-operative probabilistic DTT in determining the position of the facial nerve (relative to extrameatal portion of a vestibular schwannoma) by using the facial nerve position at surgery as a reference standard.

SECONDARY OUTCOMES:
Reproducibility | 4 years
  To assess the interobserver and intraobserver reproducibility in the assessment of cranial nerve position on pre- operative probabilistic DTT images.
Relationship of tumour size with confidence | 4 years
  To assess the relationship of tumour size with confidence when determining facial nerve position on pre-operative probabilistic DTT.
Relationship of tumour size with accuracy | 4 years
  To assess the relationship of tumour size with accuracy when determining facial nerve position on pre-operative probabilistic DTT.
Facial nerve shape | 4 years
  To compare the surgical assessment of facial nerve shape (compact or flat morphology, secondary to tumour-related pressure effects) with the ability to assess facial nerve position on pre-operative probabilistic DTT images.
Comparison of DTT with conventional anatomical sequence | 4 years
  To compare the confidence and accuracy of pre-operative probabilistic DTT with high resolution T2w imaging (a standard anatomical MRI sequence obtained on routine pre-operative scanning) when determining facial nerve position.
Assessment of adjacent CPA nerves. | 4 years
  To assess whether adjacent cranial nerves that lie at the cerebellopontine angle (base of the brain) and internal auditory meatus (inner ear canal) can be detected with pre-operative probabilistic DTT.

CONTACTS AND LOCATIONS:
Overall Officials: Steve Connor, MBBS, FRCR, Principal Investigator — King's College Hospital NHS Trust
Locations (1):
- King's College Hospital NHS Foundation Trust, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cauley KA, Filippi CG. Diffusion-tensor imaging of small nerve bundles: cranial nerves, peripheral nerves, distal spinal cord, and lumbar nerve roots--clinical applications. AJR Am J Roentgenol. 2013 Aug;201(2):W326-35. doi: 10.2214/AJR.12.9230. PMID 23883249
- [Background] Choi KS, Kim MS, Kwon HG, Jang SH, Kim OL. Preoperative identification of facial nerve in vestibular schwannomas surgery using diffusion tensor tractography. J Korean Neurosurg Soc. 2014 Jul;56(1):11-5. doi: 10.3340/jkns.2014.56.1.11. Epub 2014 Jul 31. PMID 25289119
- [Background] Gerganov VM, Giordano M, Samii M, Samii A. Diffusion tensor imaging-based fiber tracking for prediction of the position of the facial nerve in relation to large vestibular schwannomas. J Neurosurg. 2011 Dec;115(6):1087-93. doi: 10.3171/2011.7.JNS11495. Epub 2011 Aug 26. PMID 21962081
- [Background] Mukherjee P, Berman JI, Chung SW, Hess CP, Henry RG. Diffusion tensor MR imaging and fiber tractography: theoretic underpinnings. AJNR Am J Neuroradiol. 2008 Apr;29(4):632-41. doi: 10.3174/ajnr.A1051. Epub 2008 Mar 13. PMID 18339720
- [Background] Sampath P, Rini D, Long DM. Microanatomical variations in the cerebellopontine angle associated with vestibular schwannomas (acoustic neuromas): a retrospective study of 1006 consecutive cases. J Neurosurg. 2000 Jan;92(1):70-8. doi: 10.3171/jns.2000.92.1.0070. PMID 10616085
- [Background] Song F, Hou Y, Sun G, Chen X, Xu B, Huang JH, Zhang J. In vivo visualization of the facial nerve in patients with acoustic neuroma using diffusion tensor imaging-based fiber tracking. J Neurosurg. 2016 Oct;125(4):787-794. doi: 10.3171/2015.7.JNS142922. Epub 2016 Jan 1. PMID 26722859
- [Background] Taoka T, Hirabayashi H, Nakagawa H, Sakamoto M, Myochin K, Hirohashi S, Iwasaki S, Sakaki T, Kichikawa K. Displacement of the facial nerve course by vestibular schwannoma: preoperative visualization using diffusion tensor tractography. J Magn Reson Imaging. 2006 Nov;24(5):1005-10. doi: 10.1002/jmri.20725. PMID 17031835
- [Background] Zhang Y, Mao Z, Wei P, Jin Y, Ma L, Zhang J, Yu X. Preoperative Prediction of Location and Shape of Facial Nerve in Patients with Large Vestibular Schwannomas Using Diffusion Tensor Imaging-Based Fiber Tracking. World Neurosurg. 2017 Mar;99:70-78. doi: 10.1016/j.wneu.2016.11.110. Epub 2016 Nov 30. PMID 27915063
- [Background] Zolal A, Juratli TA, Podlesek D, Rieger B, Kitzler HH, Linn J, Schackert G, Sobottka SB. Probabilistic Tractography of the Cranial Nerves in Vestibular Schwannoma. World Neurosurg. 2017 Nov;107:47-53. doi: 10.1016/j.wneu.2017.07.102. Epub 2017 Jul 25. PMID 28754643